CLINICAL TRIAL: NCT03819452
Title: Impact of Vitamin D on Acute Ischemic Stroke Prognosis
Acronym: IVASTO
Status: Completed | Type: Observational
Sponsor: Abha International Private Hospital (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: Fleifel002
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Ischemic Stroke
Keywords: vitamin D; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vitamin D Level — Vitamin D level is measured upon the presentation of the case with ischemic stroke

SUMMARY:
This is a registry for all patients admitted to hospital settings with Ischemic stroke in Mansoura University Hospital. The registry will capture patients' data, investigations and vitamin D level on admission. Follow-up is taking place using MODIFIED RANKIN SCALE

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ischemic stroke not older than 48 hours

Exclusion Criteria:

* Ischemic stroke due to accidents or any trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending to hospital settings diagnosed with ischemic stroke are investigated to have low level of vitamin D
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Correlation of Vitamin D level and the Incidence of Ischemic Stroke | On admission
  Correlation Analyses between vitamin D and ischemic stroke will be applies

SECONDARY OUTCOMES:
impact of vitamin D on ischemic stroke in relationship with gender | On admission
  subgroup analyses per gender will be applied to check the difference of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed FLeifel, MD PhD, Study Director — Abha International Private Hospital
Locations (2):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt
- IQVIA, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data of study participants will be kept confidential and no intention for distribution.